CLINICAL TRIAL: NCT05765058
Title: Randomized Clinical Trial on the Efficacy of Professionally and Self-applied Fluoride Varnishes, Solutions and Mousse on Arresting Root Caries
Brief Title: The Efficacy of Tooth Mouse, SFD and NaF in Caries Activity in Root Caries. A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Arresting root caries
Record Dates: First submitted 2023-02-13; First posted 2023-03-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Root Caries; NaF; SDF; Tooth Mousse
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Intervention Model Description: RCT (Randomized Clinical Study)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Assessor do not know to which group the testing product belongs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SDF solution (Placebo Comparator): Subjects will receive one of the available non-operative treatment methods for root caries, namely silver diamine fluoride solution (SDF [38% F-, 38,000 ppm F]) twice yearly applied professionally by a dentist, Placebo Tooth mousse twice daily applied at home by the subject and will perform tooth brushing with regular fluoridated toothpaste (NaF, [0.32% F-, 1,450 ppm F]) twice daily.
  Interventions: Other: Group A
- NaF Varnish (Placebo Comparator): Subjects will receive one of the available non-operative treatment methods for root caries, namely sodium fluoride varnish (NaF, [5% F-, 22,600 ppm F]) twice yearly applied professionally by a dentist, Placebo Tooth mousse twice daily applied at home by the subject and will perform tooth brushing with regular fluoridated toothpaste (NaF, [0.32% F-, 1,450 ppm F]) toothpaste twice daily.
  Interventions: Other: Group B
- Tooth mousse (Experimental): Subjects will receive placebo varnish (water-based) twice yearly applied professionally by a dentist, Biosmalto Tooth mousse twice daily applied at home by the subject and will perform tooth brushing with regular fluoridated toothpaste (NaF, [0.32% F-, 1,450 ppm F]) toothpaste twice daily.
  Interventions: Other: Group C
- Placebo varnish (Sham Comparator): Subjects will receive placebo varnish (water-based) twice yearly applied professionally by a dentist, Placebo tooth mousse twice daily applied at home by the subject and will perform tooth brushing with regular fluoridated toothpaste (NaF, [0.32% F-, 1,450 ppm F]) toothpaste twice daily.
  Interventions: Other: Group D

INTERVENTIONS:
Other: Group A — Application of SDF (silver diamine fluoride) solution on the root caries lesions twice yearly in a professional setting. Application of Placebo tooth mousse by the subject twice daily. Regular tooth brushing with standardized fluoridated toothpaste.
  Arms: SDF solution
Other: Group B — Application of Sodium Fluoride varnish on the root caries lesions twice yearly in a professional setting. Application of Placebo tooth mousse by the subject twice daily. Regular tooth brushing with standardized fluoridated toothpaste.
  Arms: NaF Varnish
Other: Group C — Application of Placebo varnish (water-based) solution on the root caries lesions twice yearly in a professional setting. Application of Biosmalto tooth mousse by the subject twice daily. Regular tooth brushing with standardized fluoridated toothpaste.
  Arms: Tooth mousse
Other: Group D — Application of Placebo varnish (water-based) solution on the root caries lesions twice yearly in a professional setting. Application of Placebo tooth mousse by the subject twice daily. Regular tooth brushing with standardized fluoridated toothpaste.
  Arms: Placebo varnish

SUMMARY:
The aim of this study is to summarize the current level of evidence on the prevalence of root caries in elderly population, evaluate the prevalence of root caries in elderly patients living in Canton Bern, Switzerland and to analyze the association between the data collected with demographic and relevant socioeconomic factors, provide relevant long-term clinical, radiographic and oral health related outcomes and to establish a pivotal reference in treatment of elderly patients by means of non-operative root caries treatment.

DETAILED DESCRIPTION:
The study aims to systematically screen the available literature in order to investigate the global root caries prevalence in particular focusing on its correlation with the published data from Switzerland. For this specific research, a comprehensive systematic review of the literature will be conducted. The aim is to summarize the level of evidence on the oral health status of the elderly, in order to gain insights in this relevant research field. By better understanding the actual situation, existing measures focusing on the situation in Switzerland will be identified by pointing of omissions/deficiencies in order to recommend new research directions for their use in future oral health outcomes research.

Thereafter, the study will evaluate the prevalence of root caries in the elderly population living in Canton Bern, Switzerland and analyze the association between the oral data collected with demographic, socioeconomic factors and compromising health conditions. Therefore, a randomized clinical trial with participants older than 45 years limited to Canton Bern will be conducted. To be representative of Canton Bern, a sample size calculation of a total of 136 subjects (sample size calculation n=107 + 25 per cent drop-out) will be applied.

Long-term non-operative treatment results as well as the oral-health status of elderly patients (>45 years of age) having received one of the non-operative treatment methods for root caries treatment will be assessed. From the original pool of patients from Canton Bern all selected individuals will receive one of the non-operative treatment methods for root caries treatment. For the present study, only data collected from patients older than 45 years old at the time of the clinical examination will be used for analysis. The clinical appearance of each root caries lesion will be recorded longitudinally at intervals of up to 6 months and followed up to 18 months. At every single visit the lesions will be clinically and photographically characterized with respect to texture (light probing), color and surface structure (visual inspection and photographic recording) and presence or absence of plaque. If occurrence of presence of plaque and/or gingival trauma is detected, they will be accompanied by oral health instruction at every visit. All participants of the study will receive

* Regular therapy with fluoride toothpaste,
* Placebo or fluoride tooth mousse for at home-use and additionally,
* Twice-yearly professional placebo or fluoride varnish/solution application.

ELIGIBILITY:
Inclusion Criteria:

* Being resident in the area of the canton Bern,
* Age >44 years,
* Three or more root caries
* Lesions ICDAS (W1 or W2) on the first premolar, canines and front teeth of the upper and lower jaw,
* Written declaration of informed consent,
* Capacity to understand questionnaire items related to the compliance of the trial.

Exclusion Criteria:

* Living in long-term care facilities, prisons, hospitals etc.,
* Known allergic reaction to oral hygiene products and/or medication and/or dental material previously used in the mouth or pharynx,
* Inability to follow the procedures of filling out questionnaires or clinical examination, e.g. physical inability to fill in questionnaires

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Significant inactivation of root caries lesion measured by visual tactile method | 18 months
  Daily use of a regularly fluoridated toothpaste and daily use of a fluoridated tooth mouse inactivate significantly more root lesions than the daily use of a regularly fluoridated toothpaste and daily use of a placebo toothpaste
Inactivation of root caries due to regular use of fluoridated toothpaste and 6-monthly use measured by visual tactile method | 6 month to 1 year
  Daily use of a regularly fluoridated toothpaste and 6-monthly use of a fluoride solution inactivate significantly more root lesions than the daily use of a regularly fluoridated toothpaste and daily use of a placebo toothpaste
Inactivation of root caries due to regular use of fluoridated toothpaste and 6-monthly use of the fluoride varnish measured by visual tactile method | 6 months to one year
  Daily use of a regularly fluoridated toothpaste and 6-monthly use of a fluoride varnish inactivate significantly more root lesions than the daily use of a regularly fluoridated toothpaste and daily use of a placebo toothpaste

SECONDARY OUTCOMES:
Data collection of root caries prevalence (number of lesion and activity status) | 18 months
  Summary of the world-wide current level of evidence on the prevalence of root caries in elderly population in Canton Bern, focusing on the published data from Switzerland.
Long-term clinical, radiographical and oral health related outcomes (Number of teeth present in the oral cavity) for senior population suffering from root caries | 18 months
  Provision of relevant long-term clinical, radiographic and oral health related outcomes and to establish a pivotal reference in treatment of elderly patients by means of non-operative root caries treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Maklennan, Principal Investigator — University of Bern
Locations (1):
- Zahnmedizinklinik University of Bern, Department of Restorative, Preventive and Paediatric Dentistry, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No